CLINICAL TRIAL: NCT00152763
Title: Psychological Support for Patients With an Implantable Cardioverter Defibrillator
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Jane Irvine, University Health Network, Toronto General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NA 5170; Grant number NA 5170
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2011-01-28 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Anxiety; Depression
Keywords: health anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Cognitive Behavior Therapy - males (Experimental): Eight telephone sessions of cognitive behavior therapy tailored to psychological adaptation to an ICD, plus a psycho-educational booklet for participants and a therapist manual. This arm included the males.
  Interventions: Behavioral: Cognitive Behaviour Therapy (CBT)
- Cognitive Behavior Therapy - females (Experimental): Eight telephone sessions of cognitive behavior therapy tailored to psychological adaptation to an ICD, plus a psycho-educational booklet for participants and a therapist manual. This arm included the females.
  Interventions: Behavioral: Cognitive Behaviour Therapy (CBT)
- Usual Cardiac Care - Males (Active Comparator): The UCC was defined as whatever the respective ICD treatment sites routinely offer their patients. All patients received standard educational materials explaining their heart disease and the ICD device. Follow-up appointments include device interrogation (i.e., to extract arrhythmia events and ICD therapies) and trouble-shooting at 6-months intervals, cardiac care as necessary, and nonsystematic supportive reassurance delivered informally in the clinic. Each centre also had access to a cardiac rehabilitation program and psychiatric consultation as needed. This arm was just for males randomized.
  Interventions: Other: Usual Cardiac Care (UCC)
- Usual Cardiac Care - females (Active Comparator): The UCC was defined as whatever the respective ICD treatment sites routinely offer their patients. All patients received standard educational materials explaining their heart disease and the ICD device. Follow-up appointments include device interrogation (i.e., to extract arrhythmia events and ICD therapies) and trouble-shooting at 6-months intervals, cardiac care as necessary, and nonsystematic supportive reassurance delivered informally in the clinic. Each centre also had access to a cardiac rehabilitation program and psychiatric consultation as needed. This arm was for females randomized.
  Interventions: Other: Usual Cardiac Care (UCC)

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy (CBT) — Cognitive behavior therapy tailored to psychological adaptation to an ICD, included 8 telephone counselling sessions, plus psycho-educational booklet and a therapist manual.
  Arms: Cognitive Behavior Therapy - females; Cognitive Behavior Therapy - males
Other: Usual Cardiac Care (UCC) — Usual cardiac care (UCC) was defined as whatever the respective ICD treatment sites routinely offer their patients. All patients received standard educational materials explaining their heart disease and the ICD device. Follow-up appointments include device interrogation (i.e., to extract arrhythmia events and ICD therapies) and trouble-shooting at 6-months intervals, cardiac care as necessary, and nonsystematic supportive reassurance delivered informally in the clinic. Each centre also had access to a cardiac rehabilitation program and psychiatric consultation as needed.
  Arms: Usual Cardiac Care - Males; Usual Cardiac Care - females

SUMMARY:
About 30% of patients survive a cardiac arrest, and the majority of these receive an implantable cardioverter defibrillator (ICD) for prevention of sudden cardiac death (SCD). While ICD therapy offers survival benefit over drug therapy, there remain significant quality of life (QL) issues. About 50% of patients experience chronic anxiety about receiving an ICD shock. Anxiety and depression in turn appear to predispose to more arrhythmias necessitating ICD therapy. The aims of the current study are:

1. to evaluate a 8-session psychosocial intervention to help patients cope effectively with receiving an ICD for secondary prevention of SCD,
2. to determine if baseline measures of depression and anxiety predict ICD therapies (i.e., anti-tachycardia pace terminations and shocks); and
3. to explore if the psychosocial intervention results in less need for appropriate ICD therapies.

DETAILED DESCRIPTION:
About 30% of patients survive a cardiac arrest, and the majority of these receive an implantable cardioverter defibrillator (ICD) for prevention of sudden cardiac death (SCD). While ICD therapy offers survival benefit over drug therapy, there remain significant quality of life (QL) issues. About 50% of patients experience chronic anxiety about receiving an ICD shock. Anxiety and depression in turn appear to predispose to more arrhythmias necessitating ICD therapy. The aims of the current study are:

1. to evaluate a 8-session psychosocial intervention to help patients cope effectively with receiving an ICD for secondary prevention of SCD,
2. to determine if baseline measures of depression and anxiety predict ICD therapies (i.e., anti-tachycardia pace terminations and shocks); and
3. to explore if the psychosocial intervention results in less need for appropriate ICD therapies.

This study will randomize 218 ICD patients to receive either usual cardiac care (n=109) OR usual cardiac care plus CBT (n=109). Participants are recruited from two hospitals in Toronto that perform ICD implants (St. Michael's Hospital and the Toronto General Hospital). Counselling follows a CBT manual and involves both face-to-face sessions and telephone sessions. The telephone is employed as a means to deliver therapy as at least half of our ICD subjects reside outside of Toronto and all patients are prohibited from driving an automobile for the first six months following ICD implant. Outcome is assessed 6 and 12-months following the date of randomization and include measures of psychological function and quality of life. Secondary outcome is frequency of ICD therapies over follow-up (i.e., anti-tachycardia pacing terminations and DC shocks).

Inclusion Criteria:

* Patients from either Toronto General hospital or St. Michael's Hospital who have coronary heart disease,
* Receiving their first ICD implant for secondary prevention of SCD or primary prevention of SCD if their underlying heart disease was hypertrophic cardiomyopathy.

Exclusion Criteria:

* Not able to read or understand English;
* Evidence of psychosis, dementia or cognitive impairment as documented in the patients' hospital records;
* Receiving an ICD for primary prevention of ICD.

ELIGIBILITY:
Inclusion Criteria:

* Patients from either Toronto General hospital or St. Michael's Hospital who have coronary heart disease,
* Receiving their first ICD implant for secondary prevention of SCD or for primary prevention of SCD and their underlying heart disease was hypertrophic cardiomyopathy.

Exclusion Criteria:

* Not able to read or understand English;
* Evidence of psychosis, dementia or cognitive impairment as documented in the patients' hospital records;
* Receiving an ICD for primary prevention of ICD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2003-10; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Irvine, D.Phil., Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Irvine, J. Stanley, J., Ong, L., Cribbie, R., Ritvo, P., Katz, J., Dorian, P., O'Donnell, S., Harris, L., Cameron, D., Hill, A., Newman, D., Johnson, S. N., Bilanovic, A. Sears, S F. Acceptability of a Cognitive Behavior Therapy Intervention to Implantable Cardioverter Defibrillator Recipients, Journal of Cognitive Psychotherapy, 2010; 24(4) (November), 243-264.
- [Derived] Ford J, Rosman L, Wuensch K, Irvine J, Sears SF. Cognitive-Behavioral Treatment of Posttraumatic Stress in Patients With Implantable Cardioverter Defibrillators: Results From a Randomized Controlled Trial. J Trauma Stress. 2016 Aug;29(4):388-92. doi: 10.1002/jts.22111. Epub 2016 Jul 14. PMID 27415850
- [Derived] Irvine J, Firestone J, Ong L, Cribbie R, Dorian P, Harris L, Ritvo P, Katz J, Newman D, Cameron D, Johnson S, Bilanovic A, Hill A, O'Donnell S, Sears S Jr. A randomized controlled trial of cognitive behavior therapy tailored to psychological adaptation to an implantable cardioverter defibrillator. Psychosom Med. 2011 Apr;73(3):226-33. doi: 10.1097/PSY.0b013e31820afc63. Epub 2011 Feb 14. PMID 21321256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment commenced in October 2003 at Toronto General Hospital and St. Michael's Hospital in Toronto, Ontario, Canada and concluded in August 2006.
Pre-assignment Details: Upon recruitment, participants completed baseline psychological assessment prior to being randomized to the experimental intervention arm (cognitive behaviour therapy) or usual care.
Groups:
- Usual Cardiac Care - Men: Cardiac care as usual for the hospital clinic which includesstandard educational materials explaining their heart disease and the ICD device. Follow-up appointments include device interrogation (i.e., to extract arrhythmia events and ICD therapies) and trouble-shooting at 6-months intervals, cardiac care as necessary, and nonsystematic supportive reassurance delivered informally in the clinic. Each centre also had access to a cardiac rehabilitation program and psychiatric consultation as needed.
- Cognitive Behaviour Therapy - Women: Eight individual sessions of cognitive behaviour therapy delivered via telephone counselling, plus a participant psycho-educational booklet
- Usual Cardiac Care - Women: Cardiac care as usual which includes standard educational materials explaining their heart disease and the ICD device. Follow-up appointments include device interrogation (i.e., to extract arrhythmia events and ICD therapies) and trouble-shooting at 6-months intervals, cardiac care as necessary, and nonsystematic supportive reassurance delivered informally in the clinic. Each centre also had access to a cardiac rehabilitation program and psychiatric consultation as needed.
- Cognitive Therapy Group - Men: Eight sessions of individual cognitive therapy delivered via telephone plus a psycho-educational booklet.
Period: Overall Study
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Started | 77 | 19 | 20 | 77
Completed | 67 | 14 | 16 | 63
Not Completed | 10 | 5 | 4 | 14
Not completed — Death | 4 | 1 | 2 | 1
Not completed — Lost to Follow-up | 6 | 4 | 2 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men | Total
Number analyzed (Participants) | 77 | 19 | 20 | 77 | 193
Age Continuous [Mean (Standard Deviation); unit: years] | 61.29 (13.17) | 54.58 (15.75) | 55.35 (18.30) | 64.2 (13.35) | 61.68 (14.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 19 | 20 | 0 | 39
  Male | 77 | 0 | 0 | 77 | 154

OUTCOME MEASURES:

1. Primary Outcome: Hospital Anxiety and Depression Scale - Depression Scale at Baseline
Description: Psychometric scale measuring symptoms of depression, score range is 0 to 24. Scores >= 8 represent clinically elevated scores. Higher scores represent greater depressive symptoms.
Time Frame: Baseline
Population: Intention to treat analyses but data on participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 4.70 (3.41) | 7.47 (5.02) | 5.35 (3.82) | 4.12 (4.01)

2. Secondary Outcome: SF-36 Mental Component Summary Scale at Baseline
Description: Quality of life measure - mental health summary, scores range from 0 to 100 with higher scores representing better mental health.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 45.90 (13.40) | 37.44 (13.69) | 42.33 (12.43) | 49.84 (10.56)

3. Primary Outcome: Hospital Anxiety and Depression Scale - Depression Scale at 6-months Follow-up
Description: as for outcome 1
Time Frame: Six-months follow-up
Population: Intention to treat analyses but data on participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 4.21 (3.31) | 4.86 (3.25) | 5.50 (4.22) | 3.82 (3.39)

4. Secondary Outcome: SF-36 Mental Component Summary Scale at 6-months Follow-up
Description: as for outcome 2
Time Frame: Six-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 48.73 (10.34) | 43.82 (11.64) | 45.67 (10.84) | 51.32 (10.99)

5. Primary Outcome: Hospital Anxiety and Depression Scale - Depression Scale at 12-months Follow-up
Description: as for outcome 1
Time Frame: Twelve-months follow-up
Population: Intention to treat analyses but data on participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 4.52 (3.29) | 4.67 (4.19) | 5.87 (3.12) | 4.15 (3.36)

6. Primary Outcome: Hospital Anxiety and Depression Scale - Anxiety Scale at Baseline
Description: Psychometric scale measuring symptoms of anxiety,score range is 0 to 24. Scores >= 8 represent clinically elevated scores. Higher scores represent greater anxiety symptoms.
Time Frame: Baseline
Population: Intention to treat analyses but data on participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 6.53 (4.26) | 9.32 (5.50) | 7.70 (3.85) | 4.80 (3.93)

7. Primary Outcome: Hospital Anxiety and Depression Scale - Anxiety Scale at 6-months Follow-up
Description: as for outcome 6
Time Frame: Six-months follow-up
Population: Intention to treat analyses but data on participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 6.06 (3.84) | 7.28 (4.01) | 6.83 (4.67) | 4.69 (3.92)

8. Primary Outcome: Hospital Anxiety and Depression Scale - Anxiety Scale at 12-months Follow-up
Description: as for outcome 6
Time Frame: Twelve-months follow-up
Population: Intention to treat analyses but data on participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 6.06 (3.97) | 8.00 (3.70) | 7.25 (3.57) | 4.43 (3.77)

9. Primary Outcome: Impact of Events Scale-Revised - Total Score at Baseline
Description: Psychometric measure of post traumatic stress disorder symptoms, scores range from 0 to 4. A score threshold of 1.4 has been found to diagnostic of post traumatic stress disorder in war veterans. Higher scores represent greater total post traumatic stress disorder symptoms.
Time Frame: Baseline
Population: Intention to treat analysis although data for participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.81 (0.66) | 1.56 (0.99) | 1.20 (0.85) | 0.63 (0.51)

10. Secondary Outcome: SF-36 Mental Component Summary Scale at 12-months Follow-up
Description: as for outcome 2
Time Frame: Twelve-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 49.92 (10.50) | 46.26 (14.00) | 41.58 (9.02) | 51.61 (46.26)

11. Primary Outcome: Impact of Events Scale-Revised - Total Score at 6-months Follow-up
Description: as for outcome 9
Time Frame: Six-months follow-up
Population: Intention to treat analysis although data for participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.70 (0.52) | 0.76 (0.83) | 0.68 (0.64) | 0.54 (0.62)

12. Primary Outcome: Impact of Events Scale-Revised - Total Score at 12-months Follow-up
Description: as for outcome 9
Time Frame: Twelve-months follow-up
Population: Intention to treat analysis although data for participants who died over follow-up were omitted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.70 (0.64) | 0.69 (0.53) | 0.82 (0.69) | 0.46 (0.47)

13. Primary Outcome: Impact of Events Scale-Revised - Intrusiveness Scale at Baseline
Description: Psychometric measure of post traumatic stress disorder intrusiveness symptoms, scores range from 0 to 4. Higher scores represent greater post traumatic stress disorder intrusiveness symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 0.80 (0.71) | 1.53 (0.98) | 1.25 (0.95) | 0.61 (0.64)

14. Primary Outcome: Impact of Events Scale-Revised - Intrusiveness Scale at 6-months Follow-up
Description: as for outcome 13
Time Frame: Six-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 0.61 (0.52) | 0.82 (0.96) | 0.73 (0.73) | 0.56 (0.73)

15. Primary Outcome: Impact of Events Scale-Revised - Intrusiveness Scale at 12-months Follow-up
Description: as for outcome 13
Time Frame: Twelve-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 0.62 (0.62) | 0.64 (0.60) | 0.80 (0.70) | 0.42 (0.47)

16. Primary Outcome: Impact of Events Scale-Revised - Avoidance Scale at Baseline
Description: Psychometric assessment of post traumatic stress disorder avoidance symptoms, scores range from 0 to 4. Higher scores represent greater post traumatic stress disorder avoidance symptoms.
Time Frame: Baseline
Population: Intention to treat analysis although data from participants who died were omitted from analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.84 (0.62) | 1.68 (1.10) | 1.25 (0.82) | 0.64 (0.58)

17. Primary Outcome: Impact of Events Scale-Revised - Avoidance Scale at 6-months Follow-up
Description: as for outcome 16
Time Frame: Six-months follow-up
Population: Intention to treat analysis although data from participants who died were omitted from analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.86 (0.64) | 0.77 (0.87) | 0.74 (0.71) | 0.55 (0.64)

18. Primary Outcome: Impact of Events Scale-Revised - Avoidance Scale at 12-months Follow-up
Description: as for outcome 16
Time Frame: Twelve-months follow-up
Population: Intention to treat analysis although data from participants who died were omitted from analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.82 (0.74) | 0.84 (0.65) | 0.98 (0.86) | 0.57 (0.66)

19. Primary Outcome: Impact of Event Scale-Revised Hyperarousal Scale at Baseline
Description: Psychometric measure of post traumatic stress disorder hyper-arousal symptoms, scores range from 0 to 4. Higher scores represent greater post traumatic stress disorder hyperarousal symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 0.78 (0.86) | 1.40 (1.11) | 1.07 (0.98) | 0.64 (0.67)

20. Primary Outcome: Impact of Event Scale-Revised Hyperarousal Scale at 6-months Follow-up
Description: as for outcome 19
Time Frame: Six-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 0.61 (0.70) | 0.64 (0.87) | 0.56 (0.61) | 0.52 (0.70)

21. Primary Outcome: Impact of Event Scale-Revised Hyperarousal Scale at 12-months Follow-up
Description: as for outcome 19
Time Frame: Twelve-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 0.64 (0.73) | 0.57 (0.54) | 0.67 (0.70) | 0.39 (0.43)

22. Primary Outcome: Crown-Crisp Experiential Index - Phobic Anxiety Scale at Baseline
Description: Psychometric measure of phobic anxiety, scores range from 1 to 3. Higher scores represent greater phobic anxiety symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.98 (0.39) | 1.17 (0.28) | 1.23 (0.41) | 0.83 (0.33)

23. Primary Outcome: Crown-Crisp Experiential Index - Phobic Anxiety Scale at 6-months Follow-up
Description: as for outcome 22
Time Frame: Six-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.92 (0.40) | 1.04 (0.38) | 1.07 (0.36) | 0.84 (0.35)

24. Primary Outcome: Crown-Crisp Experiential Index - Phobic Anxiety Scale at 12-months Follow-up
Description: as for outcome 22
Time Frame: Twelve-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 12 | 76
units on a scale | 0.98 (0.40) | 1.13 (0.35) | 1.07 (0.40) | 0.93 (0.35)

25. Secondary Outcome: SF-36 Physical Component Summary Score at Baseline
Description: Quality of life measure of physical health, scores range from 0 to 100 with higher scores representing better physical health.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 39.19 (10.46) | 36.13 (7.06) | 37.60 (11.81) | 38.85 (10.15)

26. Secondary Outcome: SF-36 Physical Component Summary Score at 6-months Follow-up
Description: as for outcome 25
Time Frame: Six-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 42.54 (10.58) | 41.46 (12.43) | 41.22 (12.85) | 42.69 (10.06)

27. Secondary Outcome: SF-36 Physical Component Summary Score at 12-months Follow-up
Description: as for outcome 25
Time Frame: Twelve-months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Number analyzed (Participants) | 73 | 18 | 16 | 76
units on a scale | 42.65 (10.33) | 42.70 (10.44) | 42.82 (14.53) | 41.54 (11.23)

28. Secondary Outcome: Percentage of Participants Who Received ICD Therapies
Description: Percentage of participants who received ICD shocks or anti-tachycardia therapies, data extracted from participants ICD devices over follow-up.
Time Frame: 12-months follow-up
Measure: Number; unit: Percentage of participants
Groups:
- Usual Cardiac Care: Cardiac care as usual for the hospital clinic which includesstandard educational materials explaining their heart disease and the ICD device. Follow-up appointments include device interrogation (i.e., to extract arrhythmia events and ICD therapies) and trouble-shooting at 6-months intervals, cardiac care as necessary, and nonsystematic supportive reassurance delivered informally in the clinic. Each centre also had access to a cardiac rehabilitation program and psychiatric consultation as needed. This includes all men and women who received UCC.
- Cognitive Behaviour Therapy: Eight individual sessions of cognitive behaviour therapy delivered via telephone counselling, plus a participant psycho-educational booklet. These data are on men and women combined within CBT.
Arm/Group | Usual Cardiac Care | Cognitive Behaviour Therapy
Number analyzed (Participants) | 97 | 96
Percentage of participants | 30.5 | 31.9

ADVERSE EVENTS:
Description: Death was the only adverse event collected.
Arm/Group | Usual Cardiac Care - Men | Cognitive Behaviour Therapy - Women | Usual Cardiac Care - Women | Cognitive Therapy Group - Men
Serious Adverse Events (participants affected / at risk) | 4/77 | 1/19 | 2/20 | 1/77
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Cardiac Care - Men (N=77) | Cognitive Behaviour Therapy - Women (N=19) | Usual Cardiac Care - Women (N=20) | Cognitive Therapy Group - Men (N=77)
Deaths (General disorders) | 4 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No